CLINICAL TRIAL: NCT07106294
Title: Systematic Evaluation of Hyperspectral Analysis as a Predictive Marker of Preeclampsia
Brief Title: Hyperspectral Imaging for Prediction of Preeclampsia
Acronym: HIPPA
Status: Recruiting | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Anna Scholz, Principal Investigator, Heidelberg University
Other Study IDs: S-313/2025
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Preeclampsia (PE) Risk; Preeclampsia
Keywords: preeclampsia; hyperspectral imaging; EASIX; endothelial dysfunction
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (serum) samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First trimester: patients scheduled for routine first trimester ultrasound assessment
- Second trimester: patients scheduled for routine anomaly scan in second trimester

SUMMARY:
Preeclampsia is a hypertensive pregnancy disorder that can quickly lead to serious, potentially life-threatening outcomes for both the mother and the fetus. Typical features of preeclampsia are by endothelial and microvascular dysfunctionsNotably, such impairments in endothelial function may precede preeclampsia diagnosis and canpersist for years postpartum. In clinical practice, however, no predictive methods have yet been established that specifically reflect endothelial dysfunction in the context of preeclampsia.

Hyperspectral imaging represents a new and non-invasive imaging modality that allows contact-free visualization of peripheral microcirculatory dynamics and tissue perfusion. Despite its growing use in other medical fields, this technology has not yet been systematically studied to determine its predictive potential in preeclampsia.

The HIPPA project (Systematic Evaluation of Hyperspectral Analysis for Prediction of Preeclampsia) is a prospective observational study to evaluate the applicability of hyperspectral imaging as a new tool for prediction of preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia is defined by hypertension in pregnancy accompanied by any systemic end-organ dysfunction. The condition can develop rapidly and is associated with significant maternal and fetal morbidity and mortality. A key component of its underlying pathophysiology is the endothelial dysfunction, which contributes to the systemic nature of the disease and the impairment of various organ systems. Importantly, these vascular alterations may not be limited to the pregnancy period but can persist after delivery and mediate long-term cardiovascular complications. Additionally, these vascular changes seem to precede the development of preeclampsia and may contribute to its pathogenesis. Pregnancy itself is often viewed as a stress test aggravating preexisting maternal subclinical cardiovascular dysfunction. Cardiovascular disease and preeclampsia are closely linked as both entities share the same risk factors and represent risk factors for each another. Cardiac remodeling has been shown to be abnormally altered in patients with a high risk for preeclampsia in the first trimester.

Hyperspectral imaging has emerged as a potentially valuable technique for assessing peripheral microcirculation and tissue perfusion in a non-invasive and contactless manner. This imaging modality captures detailed hemodynamic data by visualizing parameters such as capillary hemoglobin oxygen saturation, tissue hemoglobin distribution, and relative tissue water content. Hyperspectral imaging has not yet been studied as predictive tool for preeclampsia before.

Given the well-documented preeclampsia-related vascular changes, the investigators suggest hyperspectral analysis as a valuable tool to predict preeclampsia. By identifying early subtle changes in microcirculatory perfusion, this method could enhance early detection and enable individualized care strategies for women at risk of developing preeclampsia.

Recently, theresearch team has explored the utility of the Endothelial Activation and Stress Index (EASIX) as a potential prognostic marker in preeclampsia. EASIX is calculated based on lactate dehydrogenase, platelet count, and creatinine and reflects systemic stress and endothelial injury, its specific relationship to microvascular health and endothelial function in pregnancy remains to be elucidated. EASIX levels were significantly increased in patients with adverse maternal and perinatal outcomes and were associated with the remaining time until delivery. The investigators hypothesize that impaired microcirculatory flow may promote pathological interactions between platelets and endothelial cells-leading to cellular damage (reflected in elevated LDH), platelet depletion via activation and microembolism, and renal impairment.

The HIPPA study (Systematic Evaluation of Hyperspectral Analysis for Prediction of Preeclampsia) is the first prospective investigation to evaluate the use of hyperspectral imaging for the prediction of preeclampsia in the first and second trimester. This study aims to assess whether the hyperspectral imaging correlates with biochemical indicators such as EASIX or markers of endothelial dysfunction. The secondary objective is to evaluate the association of hyperspectral imaging and-adverse maternal and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* age ≥ 18 years
* patient's ability to provide consent
* written informed consent
* women scheduled for a routine ultrasound scan in first or second trimester

Exclusion Criteria:

* lack of consent
* language barrier
* severe fetal chromosomal/genetic/structural anomalies known at study enrollment
* smoking in the last two hours before measurement
* diagnosis of preeclampsia at study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women scheduled for a routine ultrasound scan in first or second trimester
Sampling Method: Non-Probability Sample
Enrollment: 1430 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Preeclampsia | up to one week after delivery
Risk ratio of the preeclampsia screening | baseline

SECONDARY OUTCOMES:
Number of patients with an adverse maternal event | up to one week after delivery
Number of patients with an adverse perinatal event | up to one week after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med. Alexandra von Au, Principal Investigator — University Heidelberg
Locations (1):
- Heidelberg University Hospital, Department of Gynecology and Obstetrics, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided